CLINICAL TRIAL: NCT02421198
Title: Family Focused Community Program to Prevent Type 2 Diabetes in Peripubertal Youth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arizona (Other)
Responsible Party: Principal Investigator, Melanie Hingle, Assistant Professor, University of Arizona
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1R21DK100805-01 (NIH)
Record Dates: First submitted 2015-04-15; First posted 2015-04-20 (Estimated); Results first posted 2025-12-26 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Pediatric Obesity
Keywords: Intervention Studies
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- face-to-face (Experimental): Delivery and testing of YMCA Family Diabetes Prevention Program (YFDPP) delivered face-to-face by YMCAs over 12 weeks to children age 9-12 and one parent/guardian.
  Interventions: Behavioral: YMCA Family Diabetes Prevention Program (YFDPP)
- face-to-face + mobile hybrid (Experimental): Delivery and testing of YMCA Family Diabetes Prevention Program (YFDPP) delivered face-to-face and via a mobile platform by YMCAs over 12 weeks to children age 9-12 and one parent/guardian.
  Interventions: Behavioral: YMCA Family Diabetes Prevention Program (YFDPP)

INTERVENTIONS:
Behavioral: YMCA Family Diabetes Prevention Program (YFDPP) — 12 week, group education to promote behavioral change delivered either face-to-face or via a combination of face-to-face and mobile technologies

SUMMARY:
Over one-third of children and adolescents are overweight and nearly 1 in 5 of them are obese. Metabolic syndrome, a strong predictor of Type 2 diabetes (T2D) and cardiovascular disease (CVD), occurs in up to 44% of obese youth, foreshadowing greater prevalence and earlier onset of T2D. Without effective interventions, "diabesity" will worsen, T2D prevalence will increase, and adults will face its consequences at younger ages. Given the strong association between obesity and chronic disease risk factors in youth, the investigators contend T2D prevention (and CVD prevention) is akin to weight control and obesity prevention. The objective of the proposed project is to develop a family-centered, community-based program for T2D prevention in peripubertal (9- to 12-year-old) youth. Using participatory methods, the investigators intend to adapt the successful adult-focused YMCA Diabetes Prevention Program (YDPP) for youth and families and assess the feasibility, acceptance and adherence to the YFDPP using two delivery formats: a 12-week YMCA-based face-to-face program and a 12-week combined face-to-face plus mobile device-based program. The proposed study will test the investigators premise that delivery with technology can reduce participant perceived burden, improve adherence, and lead to improved anthropometric, behavioral and physiological outcomes. The investigators will use the resulting data to design an appropriately powered full-scale trial. The importance of the proposed study is underscored both by the statistics cited above and the recent call for proposals to translate efficacious clinical interventions into effective community programs for youth. The potential impact of the proposed intervention is great in that the program will be delivered by paraprofessionals from the community without university researchers; significant in that it targets a major public health challenge in children and includes assessment of objective behavioral and clinical data; and innovative in that it focuses on an at-risk population, takes place at a popular, accessible community venue, and uses mobile technologies to extend reach and increase engagement of youth and families with intervention content. The long-term goal is to create a scalable, replicable, and sustainable program that overcomes existing barriers to implementation and dissemination of evidence-based, research-proven diabetes prevention programs to youth and families, thereby improving population health.

DETAILED DESCRIPTION:
The investigators objective is to develop a family-centered, community-based program for T2D prevention in peripubertal (9-12-year-old) youth. Efficacious community programs for youth are not available (although promising components exist), and thus the investigators propose to adapt the successful adult-focused YMCA Diabetes Prevention Program (YDPP) for youth and families, and assess its impact on anthropometric, behavioral and physiological outcomes in support of the design (power calculation) of a full-scale trial. The proposed study will evaluate the adapted program using two formats (with and without mobile technologies). Secondary endpoints will include participant perceived burden, adherence, and program costs.

Aim 1: Adapt an efficacious diabetes prevention program in adults (the YMCA Diabetes Prevention Program, or YDPP) for delivery to overweight peripubertal youth and their families, thereby establishing a YMCA Family Diabetes Prevention Program (YFDPP).

Aim 2: Test the feasibility, participant acceptance (child and parent) and retention rates of the YFDPP using two formats, a 12-week YMCA-based face-to-face program and a 12-week program with content delivered through a combination of face-to-face and mobile devices.

Aim 3: Test the impact of the new YFDPP using two formats on anthropometric (height, weight, BMI and waist circumference), behavioral (diet and physical activity), and physiological (fasting insulin, glucose, lipid) outcomes, using the resulting data to design an appropriately powered full-scale trial.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria for Children and Parents/Primary Caregivers

* child's age between 9 to 12 years
* child body mass index (BMI) 85th percentile for age and sex
* child has T2D risk factors:

  * 1st or 2nd degree relative with T2D
  * conditions associated with insulin resistance/metabolic syndrome (e,g, acanthosis nigricans, hypertension, dyslipidemia, PCOS, or small for gestational age birth weight, maternal history of T2D or gestational diabetes)
* parent/primary caregiver must be willing to participate in intervention sessions and activities (note: primary caregiver is the adult guardian who most frequently prepares/obtains food, regulates media use, and provides physical activity opportunities for the child)
* parent/child willing to use a study-provided mobile device during intervention
* parent and child speak and read English

Exclusion Criteria:

Exclusion Criteria for Children (Index Participants) and Parents/Primary Caregivers

* child/parent unwillingness to participate in group activities or to use study-provided mobile device
* child previously diagnosed T1 or T2D
* child with psychiatric disturbances or mental illness
* child with inability to be physically active
* child/parent inability to speak and read English
* child takes weight loss medications or medications known to cause weight gain or affect appetite.

Ages: 9 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 47 (Actual)
Dates: Start 2015-05; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hingle MD, Turner T, Kutob R, Merchant N, Roe DJ, Stump C, Going SB. The EPIC Kids Study: a randomized family-focused YMCA-based intervention to prevent type 2 diabetes in at-risk youth. BMC Public Health. 2015 Dec 18;15:1253. doi: 10.1186/s12889-015-2595-3. PMID 26679186

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Face-to-face | Face-to-face + Mobile Hybrid
Started | 25 | 22
Completed | 18 | 18
Not Completed | 7 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Face-to-face | Face-to-face + Mobile Hybrid | Total
Number analyzed (Participants) | 25 | 22 | 47
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 25 | 22 | 47
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 10.8 (1.17) | 11 (1.3) | 10.9 (1.21)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 10 | 21
  Male | 14 | 12 | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 8 | 19
  Not Hispanic or Latino | 7 | 8 | 15
  Unknown or Not Reported | 7 | 6 | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 5 | 10
  White | 11 | 9 | 20
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 8 | 7 | 15
BMI z score [Mean (Standard Deviation); unit: z-score] — Scores of 0 correspond to the average BMI for age and sex. Positive z-scores indicate a BMI above the population average (higher relative weight for height), and negative z-scores indicate a BMI below the population average (lower relative weight for height). For example, a BMI z-score of +1.96 corresponds approximately to the 97.5th percentile for BMI, indicating that an individual's BMI is higher than 97.5% of age- and sex-matched peers in the reference population.
  z-score | 1.97 (0.08) | 1.96 (0.09) | 1.97 (0.37)

OUTCOME MEASURES:

1. Primary Outcome: Change in Percentage Overweight
Description: Percentage overweight will be calculated as percentage over the median body mass index (BMI) for age and gender and change in BMI zscore
Time Frame: Baseline, Week 12 (post-intervention)
Population: Pre- and post-intervention measurements for each of the 36 participating youth were used to calculate difference in chance in % overweight between those two study time points by intervention arm (n=18 in each arm).
Measure: Mean (Standard Deviation); unit: change in percent overweight
Arm/Group | Face-to-face | Face-to-face + Mobile Hybrid
Number analyzed (Participants) | 18 | 18
change in percent overweight | 1.92 (0.10) | 1.91 (0.09)

2. Secondary Outcome: Dietary Intake
Description: Diet quality was assessed using the Healthy Eating Index-2010 (HEI-2010), which measures adherence to the 2010 Dietary Guidelines for Americans. Scores range from 0 to 100, with higher scores indicating greater adherence and better diet quality.
  HEI-2010 scores were computed from 24-hour recall data collected at baseline and Week 12 (post-intervention).
Time Frame: Baseline, Week 12 (post-intervention)
Population: Thirty-seven participants who completed both baseline and Week 12 dietary recalls were included in this analysis.
Measure: Mean (Standard Deviation); unit: score (1-100)
Groups:
- Face-to-face: Delivery and testing of YMCA Family Diabetes Prevention Program (YFDPP) delivered face-to-face by YMCAs over 12 weeks to children age 9-12 and one parent/guardian.
  YMCA Family Diabetes Prevention Program(YFDPP): 12 week, group education to promote behavioral change delivered either face-to-face or via a combination of face-to-face and mobile technologies
- Face-to-face + Mobile Hybrid: Delivery and testing of YMCA Family Diabetes Prevention Program (YFDPP) delivered face-to-face and via a mobile platform by YMCAs over 12 weeks to children age 9-12 and one parent/guardian.
  YMCA Family Diabetes Prevention Program(YFDPP): 12 week, group education to promote behavioral change delivered either face-to-face or via a combination of face-to-face and mobile technologies
Arm/Group | Face-to-face | Face-to-face + Mobile Hybrid
Number analyzed (Participants) | 24 | 13
score (1-100)
  Baseline | 48.6 (9) | 47.7 (9.5)
  Week 12 | 47.8 (9.4) | 51.4 (10.2)

3. Secondary Outcome: Physical Activity
Description: Physical activity was objectively measured using GT3X accelerometers worn on the hip for 7 consecutive days at baseline and again at Week 12 (post-intervention). Data were processed using ActiLife software with standard youth cut points to classify activity intensity levels.
Time Frame: Baseline, Week 12 (post-intervention)
Population: Thirty-three participants who provided valid accelerometer data (≥4 days of wear time, ≥10 hours per day) at both baseline and Week 12 were included in this analysis.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Face-to-face | Face-to-face + Mobile Hybrid
Number analyzed (Participants) | 20 | 13
minutes
  Baseline | 22.6 (11.1) | 35.8 (16.6)
  Week 12 | 27.8 (20) | 33.5 (17.4)

4. Secondary Outcome: Change in Waist Circumference
Description: Waist circumference (cm) was measured at the level of the umbilicus using a non-stretchable measuring tape, following standard anthropometric procedures. Measurements were taken at baseline and at Week 12 (post-intervention) with participants standing and breathing normally.
  The reported value represents the mean change in waist circumference from baseline to Week 12 across all participants. The change score was calculated as the Week 12 measurement minus the baseline measurement; positive values indicate an increase and negative values indicate a decrease in waist circumference over the 12-week intervention period.
Time Frame: Baseline, Week 12 (post-intervention)
Measure: Mean (95% Confidence Interval); unit: cm
Groups:
- Face-to-face + Mobile Hybrid: Delivery and testing of YMCA Family Diabetes Prevention Program (YFDPP) delivered face-to-face and via a mobile platform by YMCAs over12 weeks to children age 9-12 and one parent/guardian.
  YMCA Family Diabetes Prevention Program(YFDPP): 12 week, group education to promote behavioral change delivered either face-to-face or via a combination of face-to-face and mobile technologies
Arm/Group | Face-to-face | Face-to-face + Mobile Hybrid
Number analyzed (Participants) | 18 | 18
cm | 0.25 [-8.61 to 9.11] | -1.15 [-15.68 to 13.37]

5. Other Pre Specified Outcome: Fasting Lipids
Description: Total cholesterol (mg/dL) was measured from fasting venous blood samples collected at baseline and Week 12 (post-intervention). The reported value represents the mean change in fasting total cholesterol from baseline to Week 12 across all participants. The change score was calculated as the Week 12 value minus the baseline value for each participant; positive values indicate an increase and negative values indicate a decrease in total cholesterol during the 12-week intervention period.
  Because this was a feasibility study not powered to detect between-group differences, results for both delivery formats (face-to-face and hybrid) were analyzed in aggregate. Arm-level estimates were not calculated or retained, as separate estimates were not meaningful for this exploratory outcome.
Time Frame: Baseline, Week 12 (post-intervention)
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Fasting Glucose
Description: Fasting plasma glucose (mg/dL) was measured from venous blood samples collected after an overnight fast at baseline and at Week 12 (post-intervention). The reported value represents the mean change in fasting glucose from baseline to Week 12 for all participants combined. The change score was calculated as the Week 12 value minus the baseline value for each participant; positive values indicate an increase and negative values indicate a decrease in fasting glucose during the 12-week intervention period.
  Because this was a feasibility study not powered for between-group comparisons, data from both intervention formats (face-to-face and hybrid) were analyzed in aggregate. Arm-level results were not calculated or retained, as separate estimates were not meaningful for this exploratory outcome.
Time Frame: Baseline and 12 week (post-intervention)
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Fasting Insulin
Description: Fasting insulin (µU/mL) was measured from venous blood samples collected after an overnight fast at baseline and at Week 12 (post-intervention). The reported value represents the mean change in fasting insulin from baseline to Week 12 for all participants combined. The change score was calculated as the Week 12 value minus the baseline value for each participant; positive values indicate an increase in fasting insulin over the 12-week intervention period, and negative values indicate a decrease. Because this was a feasibility study not powered for between-group comparisons, results were analyzed in aggregate across both intervention arms.
Time Frame: Baseline, Week 12 (post-intervention)
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Blood Pressure
Description: Blood pressure was measured in duplicate after 5 minutes of seated rest using an automated oscillometric device. The mean of the two readings was used. Because the study was designed to assess feasibility and not efficacy, blood pressure change was analyzed descriptively across the combined cohort.
Time Frame: Baseline, Week 12 (post-intervention)
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Participants were monitoring during the time they participated in the study: 6 months (12 week intervention + 14-week follow-up)
Description: The definition of adverse and/or serious adverse event does not differ than the clinicaltrials.gov definition.
Arm/Group | Face-to-face | Face-to-face + Mobile Hybrid
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/22
Other Adverse Events (participants affected / at risk) | 0/25 | 0/22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No